CLINICAL TRIAL: NCT00866515
Title: A Double-blind, Placebo-controlled, Randomised, 2-way Crossover Drug Interaction Study to Investigate the Pharmacokinetic and Pharmacodynamic Effects Following Co-administration of GW642444M With Ketoconazole
Brief Title: Drug Interaction Study to Investigate Co-administration of GW642444M With Ketoconazole
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 112205
Record Dates: First submitted 2009-01-22; First posted 2009-03-20 (Estimated); Last update posted 2017-07-18 (Actual); Status verified 2017-07

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Healthy volunteer; pharmacodynamics; Ketoconazole; Drug Interaction; pharmacokinetcs; GW642444M; pharmacokinetics
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Ketoconazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active (Experimental): Ketoconazole 400mg OD days 1-6
  Interventions: Drug: Ketoconazole + GW642444M
- Placebo (Placebo Comparator): Placebo OD for 1 to 6 days
  Interventions: Drug: Placebo + GW642444M

INTERVENTIONS:
Drug: Ketoconazole + GW642444M — Ketoconazole 400mg OD days 1-6, GW642444M 25ug single dose on D5
  Arms: Active
Drug: Placebo + GW642444M — Placebo to match D1-6 + GW642444M 25ug single dose on D5
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
This will be a single-centre, randomised, double blind, placebo controlled, two-way crossover study in healthy male and female subjects. There will be two treatment periods each consisting of 7 days. During each treatment period subjects will receive single doses of ketoconazole or placebo on the morning of days 1-6 with a single dose of GW642444M on the morning of Day 5.

DETAILED DESCRIPTION:
This will be a single-centre, randomised, double blind, placebo controlled, two-way crossover study in healthy male and female subjects. There will be two treatment periods each consisting of 7 days. During each treatment period subjects will receive single doses of ketoconazole or placebo on the morning of days 1-6 with a single dose of GW642444M on the morning of Day 5.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included at the discretion of the Investigator only if the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* AST, ALT, alkaline phosphatase and bilirubin ≤ 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Male or female between 18 and 65 years of age inclusive, at the time of signing the informed consent.
* A female subject is eligible to participate if she is of:
* Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation, hysterectomy or bilateral oophorectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 MlU/ml and estradiol < 40 pg/ml (<140 pmol/L) is confirmatory]. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the contraception methods in Section 8.1 if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrolment. For most forms of HRT, at least 2-4 weeks will elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their post-menopausal status, they can resume use of HRT during the study without use of a contraceptive method.
* Child-bearing potential and agrees to use one of the contraception methods listed in Section 8.1 for an appropriate period of time (as determined by the product label or investigator) prior to the start of dosing to sufficiently minimize the risk of pregnancy at that point. Female subjects must agree to use contraception until after the final follow-up visit has been completed.
* Body weight ≥ 50 kg and BMI within the range 19 - 29.9 kg/m2 (inclusive).
* Demonstrated ability to use the inhaler device in a satisfactory and repeatable manner
* Subjects who are current non-smokers, who have not used any inhaled tobacco products (snuff is permitted) in the 12 month period preceding the screening visit and who have a pack history of ≤ 10 pack years.
* No significant abnormality on 12-lead ECG at screening, including the following requirements:
* Ventricular rate ≥ 40 beats per minute
* PR interval ≥ 120 and ≤ 210 msec
* Q waves < 30 msec (up to 50 msec permitted in lead III only)
* QRS interval to be ≥ 60 msec and ≤ 120 msec
* QTc interval must be < 450 msec (QTcB or QTcF; machine or manual reading) based on an average from three ECGs obtained over a brief recording period
* FEV1 ≥ 80% predicted and a FEV1 / FVC ratio ≥ 0.7 at screening
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria:

* As a result of medical interview, physical examination or screening investigations, the principle investigator or delegate physician deems the subject unsuitable for the study.
* Systolic blood pressure which is outside the range 90 to 140 mmHg, diastolic blood pressure outside the range 50 to 90 mmHg or heart rate outside the range 40 to 90 bpm.
* The subject has been treated for or diagnosed with depression within six months of screening or has a history of significant psychiatric illness.
* The subject has any history of breathing problems in adult life (i.e. history of asthmatic symptomatology).
* A clinically significant abnormality on standard pulmonary function testing, or any other finding that would prevent satisfactory administration of the inhaled study medication.
* Any contraindication to the administration of ketoconazole, as described in the current [NIZORAL Product Information, Janssen-Cilag Pty Limited, 2008].
* History of sensitivity to any of the study medications, or components thereof (including milk protein) or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Currently taking regular (or a course of) medication whether prescribed or not, with the exception of those permitted medications listed in Section 8.1 and Section 9.1.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of regular alcohol consumption within 6 months of the study defined as:
* An average weekly intake of >21 units for males or >14 units for females. One unit is equivalent to 8 g of alcohol: a half-pint (~250 mL) of beer, 1 glass (100 mL) of wine or 1 measure (30 mL) of spirits.
* The subject has participated in a clinical trial and has received a drug or a new chemical entity within 30 days or 5 half-lives, or twice the duration of the biological effect of any drug (whichever is longer) prior to the first dose of current study medication.
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* The subject has donated a unit of blood within the previous 16 weeks or intends to donate within 16 weeks after completing the study.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* The subject has tested positive for HIV antibodies.
* The subject has a positive pre-study urine drug screen/ alcohol breath test. A minimum list of drugs that will be screened for include Amphetamines, Barbiturates, Cocaine, Opiates, Cannabinoids and Benzodiazepines.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subjects who have a screening haemoglobin value < 110 mg/L.
* Pregnant (as determined by positive (serum or urine) hCG test at screening or prior to dosing) or lactating females.
* Subject is mentally or legally incapacitated.
* CO breath monitoring indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
* Consumption of red wine, seville oranges, grapefruit or grapefruit juice and/or pummelos, exotic citrus fruits, grapefruit hybrids or fruit juices from 7 days prior to the first dose of study medication.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-12-22 (Actual); Primary Completion 2009-03-27 (Actual); Study Completion 2009-03-27 (Actual)

PRIMARY OUTCOMES:
Supine heart rate and blood potassium levels | Day 5

SECONDARY OUTCOMES:
Plasma GW642444M concentrations | Day 5
Reported Adverse Events | treatment periods

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Randwick, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Kempsford R, Allen A, Bal J, Rubin D, Tombs L. The effect of ketoconazole on the pharmacokinetics and pharmacodynamics of inhaled fluticasone furoate and vilanterol trifenatate in healthy subjects. Br J Clin Pharmacol. 2013 Jun;75(6):1478-87. doi: 10.1111/bcp.12019. PMID 23116485
- See also: Results for study 112205 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/112205?search=study&search_terms=112205#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: 112205 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 112205 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 112205 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 112205 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 112205 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 112205 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 112205 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register